CLINICAL TRIAL: NCT00546169
Title: Non-interventional Trial About Treatment of Haemorrhages in Cholecystectomy With TachoSil (TC-027-DE)
Status: Completed | Type: Observational
Sponsor: Nycomed (Industry)
Responsible Party: Nycomed, Clinical Trial Operations
Other Study IDs: TC-027-DE
Record Dates: First submitted 2007-10-17; First posted 2007-10-18 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2008-08

CONDITIONS: Hemorrhage
Keywords: Patients undergoing elective or acute cholecystectomy
MeSH Terms: conditions — Hemorrhage | interventions — Fibrinogen; Thrombin; TachoSil

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A
  Interventions: Drug: Fibrinogen (human) + thrombin (human) (TachoSil)

INTERVENTIONS:
Drug: Fibrinogen (human) + thrombin (human) (TachoSil) — haemorrhages in cholecystectomy

SUMMARY:
* Effectiveness and reliability of TachoSil in cholecystectomy (elective and acute)
* Evaluation of TachoSil in laparoscopic cholecystectomy
* Risk profile of patient under anticoagulant therapy undergoing acute cholecystectomy
* Pharmaco-economic evaluation
* Recording of AE's/SAE's Considering the total number of cholecystectomies in Germany (170.000 cases/y), out of them about 75% laparoscopic and 10.000 conversions totally it seems urgent to record data about usage of TachoSil in such procedures. For the time being TachoSil is applied in about 2% of the gall bladder procedures.

Aim is to evaluate a possible patient and procedure profile where TachoSil is most beneficial.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective or acute cholecystectomy
* The only restrictions of use will be those resulting from the contraindications (see section 4.3 of the Summary of Product Characteristics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: care clinic
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nycomed Clinical Trial Operations, Study Chair — Headquaters
Locations (1):
- Nycomed, Roskilde, Denmark